CLINICAL TRIAL: NCT00667654
Title: A Phase 2, Open-label Study to Evaluate Safety and Tolerability, and to Explore the Efficacy, of Dosing Regimens of Intraarticular 4975 in Patients With Chronic Moderate to Severe Pain of the Knee Associated With Osteoarthritis
Brief Title: Safety and Tolerability of 4975 in the Treatment of Moderate to Severe Knee Pain Due to Osteoarthritis (OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114-02P
Record Dates: First submitted 2008-04-23; First posted 2008-04-28 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — CNTX-4975

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 100-200 µg CNTX-4975 (Experimental): single dose
  Interventions: Drug: CNTX-4975
- 300-425 µg CNTX-4975 (Experimental): Total dose delivered as two separate lower doses
  Interventions: Drug: CNTX-4975
- 600-700 µg CNTX-4975 (Experimental): Total dose delivered as two separate lower doses
  Interventions: Drug: CNTX-4975
- 800 µg CNTX-4975 (Experimental): Total dose delivered as two separate lower doses
  Interventions: Drug: CNTX-4975
- 900-1000 µg CNTX-4975 (Experimental): Total dose delivered as two separate lower doses
  Interventions: Drug: CNTX-4975

INTERVENTIONS:
Drug: CNTX-4975 — Testing a range of dosing configurations to optimize patient tolerability

SUMMARY:
This study will evaluate dosing regimens of 4975 in terms of safety and tolerability when delivered as an intra-articular injection in the knee. Secondary objectives will be to explore the efficacy of 4975 in terms of onset, extent and duration of pain relief.

DETAILED DESCRIPTION:
This is a single site study. The study drug, 4975, will be administered in various dosing regimens by intra-articular injection followed by an observation period of up to 12 weeks. Pain in the treated knee will be assessed before, during and after administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 40 years or over.
* Body mass index (BMI) of 35 or less.
* History of OA of the knee for at least 1 year and has experienced pain in the target area for at least six months.
* X-Ray of the target knee.
* Willing and able to complete the study procedures.

Exclusion Criteria:

* Female patients who are pregnant or lactating or who plan to get pregnant.
* Clinically significant form of joint disease other than OA.
* Medical condition that could adversely impact the patient's participation, safety or affect the conduct of the study.
* Prior major trauma in the target knee or major surgeries such as partial or total knee arthroplasty.
* Arthroscopic surgery on the target knee within 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of IA CNTX-4975 as measured by related AEs occurring on day of dosing measures of pain at prescribed times | 12 Weeks

SECONDARY OUTCOMES:
Evaluate analgesic efficacy, as measured by the PGIC, following IA injection of CNTX-4975 | 12 Weeks
Change from baseline to Week 12 in WOMAC subscale score | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William C Houghton, MD, Study Director — Anesiva, Inc.; Shaun Comfort, MD, MBA, Study Director — Anesiva, Inc.
Locations (1):
- Clinical Phamacology Study Group, Worcester, Massachusetts, United States